CLINICAL TRIAL: NCT07039916
Title: A Phase 3, Multicenter, Randomized, Placebo-Controlled, Double-Blind Study to Assess the Efficacy and Safety of IMVT-1402 in Patients With Mild to Severe Generalized Myasthenia Gravis
Brief Title: Study to Assess the Efficacy and Safety of IMVT-1402 in Participants With Mild to Severe Generalized Myasthenia Gravis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Immunovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IMVT-1402-3101; 2024-515979-35-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Generalized Myasthenia Gravis
Keywords: IMVT-1402; Generalized Myasthenia Gravis; Acetylcholine receptor; Muscle-specific kinase; Autoantibody; Lipoprotein receptor-related protein 4; Autoimmune disease; Neonatal fragment crystallizable receptor (FcRn)
MeSH Terms: conditions — Myasthenia Gravis; Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The Sponsor will also be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: IMVT-1402 Dose 1 (Experimental)
  Interventions: Drug: IMVT-1402
- Group 2: IMVT-1402 Dose 2 (Experimental)
  Interventions: Drug: IMVT-1402
- Placebo/ IMVT-1402 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: IMVT-1402

INTERVENTIONS:
Drug: IMVT-1402 — • Dose 1 subcutaneous (SC) once weekly (QW) for 12 weeks (Period 1)
  Arms: Group 1: IMVT-1402 Dose 1
Drug: IMVT-1402 — * Dose 2 SC QW for 12 weeks (Period 1)
  * Dose 2 SC QW for 14 weeks (Period 2)
  * Dose 2 SC QW for 52 weeks (Period 3)
  Arms: Group 2: IMVT-1402 Dose 2
Drug: Placebo — • Placebo SC QW for 12 weeks (Period 1)
  Arms: Placebo/ IMVT-1402
Drug: IMVT-1402 — * Dose 1 SC QW for 14 weeks (Period 2)
  * Dose 1 SC QW for 52 weeks (Period 3)
  Arms: Group 1: IMVT-1402 Dose 1; Placebo/ IMVT-1402

SUMMARY:
The purpose of the study is to assess the efficacy, safety and tolerability of IMVT-1402 in adult participants with mild to severe generalized myasthenia gravis.

ELIGIBILITY:
Inclusion Criteria:

* Participants with the ability to understand the requirements of the trial, provide written informed consent, and comply with the trial protocol procedures.
* Have mild to severe gMG by Myasthenia Gravis Foundation of America (MGFA) classification of Class II, III, or IVa at the Screening Visit
* Have an MG activities of daily living (MG-ADL) score of ≥ 6 at the Screening Visit and Baseline Visit (Day 1)

Additional inclusion criteria are defined in the protocol.

Exclusion Criteria:

* Have experienced myasthenic crisis within 12 weeks prior to the Screening Visit.
* Have had a thymectomy performed < 6 months prior to the Screening Visit or have a planned thymectomy during the study
* Have any active or untreated malignant thymoma

Additional exclusion criteria are defined in the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in MG-ADL Score for Antibody-positive Participants | Baseline to Week 12

SECONDARY OUTCOMES:
Change from Baseline in Quantitative Myasthenia Gravis (QMG) Score for Antibody-positive Participants | Baseline to Week 12
Percentage of Antibody-positive Participants Achieving MG-ADL Score of 0 or 1 | Week 12
Percentage of Antibody-positive Participants with ≥50% Improvement in MG-ADL Score | Baseline to Week 12

CONTACTS AND LOCATIONS:
Locations (58):
- United States (38):
  - Site Number - 1041, Mobile, Alabama
  - Site Number - 1017, Phoenix, Arizona
  - Site Number - 1025, Scottsdale, Arizona
  - Site Number - 1042, Tucson, Arizona
  - Site Number - 1010, Carlsbad, California
  - Site Number - 1028, Irvine, California
  - Site Number - 1023, Los Angeles, California
  - Site Number - 1029, Rancho Mirage, California
  - Site Number - 1004, San Francisco, California
  - Site Number - 1027, Fort Collins, Colorado
  - Site Number - 1001, New Haven, Connecticut
  - Site Number - 1024, Washington D.C., District of Columbia
  - Site Number - 1006, Clearwater, Florida
  - Site Number - 1037, Ormond Beach, Florida
  - Site Number - 1002, Port Charlotte, Florida
  - Site Number - 1050, Rockledge, Florida
  - Site Number - 1007, Tampa, Florida
  - Site Number - 1014, Atlanta, Georgia
  - Site Number - 1022, Lexington, Kentucky
  - Site Number - 1032, Nicholasville, Kentucky
  - Site Number - 1005, East Lansing, Michigan
  - Site Number - 1019, Totowa, New Jersey
  - Site Number - 1036, New York, New York
  - Site Number - 1034, New York, New York
  - Site Number - 1020, Chapel Hill, North Carolina
  - Site Number - 1013, Durham, North Carolina
  - Site Number - 1044, Raleigh, North Carolina
  - Site Number - 1038, Cincinnati, Ohio
  - Site Number - 1011, Yukon, Oklahoma
  - Site Number - 1031, Eugene, Oregon
  - Site Number - 1030, Charleston, South Carolina
  - Site Number - 1015, Charleston, South Carolina
  - Site Number - 1021, Memphis, Tennessee
  - Site Number - 1003, Dallas, Texas
  - Site Number - 1047, Denton, Texas
  - Site Number - 1048, Lubbock, Texas
  - Site Number - 1009, Charlottesville, Virginia
  - Site Number - 1040, Richmond, Virginia
- Site Number - 3201, Brno, Czechia
- Site Number - 3601, Copenhagen, Denmark
- Georgia (3):
  - Site Number - 8002, Tbilisi
  - Site Number - 8003, Tbilisi
  - Site Number - 8001, Tbilisi
- Germany (3):
  - Site Number - 6502, Bochum
  - Site Number - 6504, Goettigen
  - Site Number - 6503, Würzburg
- Hungary (3):
  - Site Number - 7552, Budapest
  - Site Number - 7553, Budapest
  - Site Number - 7551, Kistarcsa
- Italy (3):
  - Site Number - 6003, Bergamo
  - Site Number - 6002, Milan
  - Site Number - 6004, Rome
- Romania (2):
  - Site Number - 7502, Constanța
  - Site Number - 7501, Târgu Mureş
- Serbia (2):
  - Site Number - 9001, Belgrade
  - Site Number - 9002, Niš
- Site Number - 7103, Barcelona, Spain
- Site Number - 7002, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No